CLINICAL TRIAL: NCT00828568
Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Therapeutic Equivalence Study of Two Imiquimod Cream 5% Treatments for Patients With Actinic Keratosis
Brief Title: Bioequivalence Study of Two Imiquimod Cream 5%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIQ-0403
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2013-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Imiquimod 5% Taro (Experimental): Imiquimod 5% manufactured by Taro applied for 16 weeks
  Interventions: Drug: Imiquimod 5% manufactured by Taro
- Aldara - Imiquimod 5% (Active Comparator): Aldara, Imiquimod 5% applied for 16 weeks
  Interventions: Drug: Aldara - Imiquimod 5%
- Vehicle (Placebo Comparator): Imiquimod vehicle applied for 16 weeks
  Interventions: Drug: Imiquimod Vehicle manufactured by Taro

INTERVENTIONS:
Drug: Imiquimod 5% manufactured by Taro — Treatment applied as a thin layer to target area once a day, 2 days each week, for 16 weeks
  Arms: Imiquimod 5% Taro
Drug: Aldara - Imiquimod 5% — Treatment applied as a thin layer to target area once a day, 2 days each week, for 16 weeks
  Arms: Aldara - Imiquimod 5%
Drug: Imiquimod Vehicle manufactured by Taro — Treatment applied as a thin layer to target area once daily, 2 days each week, for 16 weeks
  Arms: Vehicle

SUMMARY:
The primary objectives are to establish the therapeutic equivalence of imiquimod cream 5%, manufactured by Taro Pharmaceuticals Inc. and Aldara (imiquimod) cream, manufactured by 3M, and to show superiority over vehicle in the treatment of AK.

The secondary objective is to compare the adverse event (AE) profiles of the two creams.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have 4 to 8 clinically diagnosed, non-hyperkeratotic, non-hypertrophic AK lesions within a 25 cm2 contiguous treatment area on either the face or balding scalp
* Women either must be 1 year post-menopausal, surgically sterile, or agree to use a medically accepted form or birth control
* Free of any systemic or dermatological disorder
* Any skin type or race, providing the skin pigmentation will allow discernment of erythema

Exclusion Criteria:

* Basal cell or squamous cell carcinoma, or other possible confounding skin conditions (on face and scalp)
* History of cutaneous hyperreactivity or facial irritation to topical products
* Engaging in activities involving excessive or prolonged exposure to sunlight
* Receiving systemic cancer chemotherapy, psoralen plus UVA therapy, UVB therapy, laser abrasion, dermabrasion, glycolic acids, or chemical peels 6 months prior to study entry
* Currently using or have used systemic steroids 2 months prior to study
* Currently using or have used on the treatment area over-the-counter retinol products, corticosteroids, cryosurgery, curettage, 5-fluorouracil, or other topical actinic keratosis treatments 28 days prior to randomization
* Pregnant or nursing mothers
* History of allergy or sensitivity to imiquimod or related compounds or other components of the formulation
* Taking immunosuppressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Investigator Site, Gilbert, Arizona
  - Investigator Site, Tempe, Arizona
  - Investigator Site, Tuscon, Arizona
  - Investigator Site, Denver, Colorado
  - Investigator Site, Jacksonville, Florida
  - Investigator Site, Miami, Florida
  - Investigator Site, Evansvill, Indiana
  - Investigator Site, Plainfield, Indiana
  - Investigator Site, Olathe, Kansas
  - Investigator Site, Wichita, Kansas
  - Investigator Site, Omaha, Nebraska
  - Investigator Site, Henderson, Nevada
  - Investigator Site, Cary, North Carolina
  - Investigator Site, Hickory, North Carolina
  - Investigator Site, High Point, North Carolina
  - Investigator Site, Winston-Salem, North Carolina
  - Investigator Site, Simpsonville, South Carolina
  - Investigator Site, Murfreesboro, Tennessee
  - Investigator Site, College Station, Texas
  - Investigator Site, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 20 dermatology clinical practices.
Groups:
- Vehicle: Patients receiving imiquimod Vehicle for 16 weeks
Period: Randomized
Arm/Group | Imiquimod 5% Taro | Aldara - Imiquimod 5% | Vehicle
Started | 184 | 179 | 62
Completed | 183 | 179 | 60
Not Completed | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Period: Treated - Received at Least One Dose
Arm/Group | Imiquimod 5% Taro | Aldara - Imiquimod 5% | Vehicle
Started | 183 | 179 | 60
Completed | 153 | 150 | 55
Not Completed | 30 | 29 | 5
Not completed — Adverse Event | 11 | 8 | 1
Not completed — Withdrawal by Subject | 9 | 11 | 0
Not completed — Lost to Follow-up | 1 | 5 | 1
Not completed — Protocol Violation | 9 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imiquimod 5% Taro | Aldara - Imiquimod 5% | Vehicle | Total
Number analyzed (Participants) | 183 | 179 | 60 | 422
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 71 | 73 | 27 | 171
  >=65 years | 112 | 106 | 33 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.5) | 67.2 (10.1) | 64.7 (9.7) | 67.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 8 | 75
  Male | 149 | 146 | 52 | 347
Region of Enrollment [Number; unit: participants]
  United States | 183 | 179 | 60 | 422

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 100% Clearance of Actinic Keratosis Lesions: Comparison of Taro Imiquimod 5% and Aldara-Imiquimod 5%
Description: Uses per protocol (PP) population.
  Each patient is assessed at 24 weeks. Actinic keratosis (AK) lesions that were identified and measured at baseline are reevaluated at the conclusion of the study. If all lesions that were identified at baseline are no longer present and there are no new lesions, the patient is 100% clear of AK lesions.
Time Frame: 24 weeks
Population: Per Protocol (PP) population
Measure: Number; unit: Participants
Arm/Group | Imiquimod 5% Taro | Aldara - Imiquimod 5%
Number analyzed (Participants) | 146 | 141
Participants | 63 | 54
Statistical Analysis 1: Comparison: Imiquimod 5% Taro vs Aldara - Imiquimod 5%; Test type: Non-Inferiority or Equivalence — The 90% confidence limit around the difference in proportion of patients considered a Treatment Success between test and reference products was calculated using Blackwelder's method with Yate's continuity correction. If the 90% confidence interval for the test to reference ratio for the primary endpoint was within -0.20 to +0.20, then the test product would have been declared therapeutically equivalent to the reference product; Mean Difference (Final Values) = 4.85, 90% CI [-5.37 to 15.08]

2. Secondary Outcome: Patients Reporting at Least One Adverse Event
Description: For all patients who received a single dose, adverse events were collected at each follow-up visit. Any patient reporting a single or multiple adverse events at any visit was conisdered to have had at least one adverse event.
Time Frame: 24 weeks
Population: Safety group includes all patients who received a single dose
Measure: Number; unit: Participants
Arm/Group | Imiquimod 5% Taro | Aldara - Imiquimod 5% | Vehicle
Number analyzed (Participants) | 183 | 179 | 60
Participants | 69 | 57 | 15

3. Primary Outcome: Number of Participants in Intention-to-treat (ITT)Population With 100% Clearance of Actinic Keratosis (AK) Lesions Identified at Baseline
Description: Uses ITT population. Three patients (1 Imiquimod 5% Taro and 2 Imiquimod Aldara) did not have a follow-up visit after dosing and were excluded from ITT. Three patients (2 Imiquimod 5% Taro and 1 Imiquimod Aldara) were not evaluable at the 24-week visit and were not in the analysis.
  Each patient is assessed at 24 weeks. Actinic keratosis (AK) lesions that were identified and measured at baseline are reevaluated at the conclusion of the study. If all lesions that were identified at baseline are no longer present and there are no new lesions, the patient is 100% clear of AK lesions.
Time Frame: 24 weeks
Population: Intention to Treat (ITT) Population
Measure: Number; unit: Participants
Arm/Group | Imiquimod 5% Taro | Aldara - Imiquimod 5% | Vehicle
Number analyzed (Participants) | 180 | 176 | 60
Participants | 74 | 64 | 6
Statistical Analysis 1: Comparison: Imiquimod 5% Taro vs Vehicle; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Aldara - Imiquimod 5% vs Vehicle; Test type: Superiority or Other; p < .0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Assessed at 24 weeks
Arm/Group | Imiquimod 5% Taro | Aldara - Imiquimod 5% | Vehicle
Serious Adverse Events (participants affected / at risk) | 4/183 | 6/179 | 1/60
Other Adverse Events (participants affected / at risk) | 22/183 | 22/179 | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod 5% Taro (N=183) | Aldara - Imiquimod 5% (N=179) | Vehicle (N=60)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod 5% Taro (N=183) | Aldara - Imiquimod 5% (N=179) | Vehicle (N=60)
APPLICATION SITE ERYTHEMA (General disorders) | 11 (12) | 8 (8) | 0 (0)
APPLICATION SITE IRRITATION (General disorders) | 5 (5) | 9 (9) | 0 (0)
APPLICATION SITE PRURITUS (General disorders) | 9 (9) | 9 (9) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days